CLINICAL TRIAL: NCT04215835
Title: Letrozole Pretreatment With Misoprostol for Induction of Abortion In First-Trimester Missed Miscarriage Among Women With One or More Previous Cesarean Deliveries.: A Randomized Controlled Trial
Brief Title: Letrozole Pretreatment With Misoprostol Induction of Abortion In First-Trimester Missed Miscarriage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: letrozole pretreatment
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Missed Abortion
MeSH Terms: conditions — Abortion, Missed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): 3 tablets of Letrozole 2.5 mg will be given as single daily dose, 7.5 mg per day for two days at home and the third dose will be given on admission to hospital on day 3 and will be followed by vaginal misoprostol 800 mcg every three hours up to maximum two doses.
  Interventions: Drug: letrozole then misoprostol
- control group (Placebo Comparator): three tablets of placebo will be given as a single daily dose, for two days at home and will be admitted on day 3 and continue treatment with misoprostol 800 mcg every three hours up to maximum two doses
  Interventions: Drug: placebo then misoprostol

INTERVENTIONS:
Drug: letrozole then misoprostol — Drug: Letrozole 2.5mg total dose 7.5 mg per day for 3 days
  Drug: Misoprostol Misoprosrol 800mcg will be given to all patients for induction of abortion
  Arms: study group
Drug: placebo then misoprostol — Drug: Placebo placebo for 3 days
  Drug: Misoprostol Misoprosrol 800mcg will be given to all patients for induction of abortion
  Arms: control group

SUMMARY:
This study compares the success rate of letrozole and misoprostol versus misoprostol alone for medical termination of first-trimester pregnancy among women with one or more previous cesarean deliveries.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age less than 64 days gestation (<9 wks).
* Hemoglobin >10 g/dL.
* BMI between 18.5 kg/m2 and 25 kg/m2.
* Missed abortion.
* previous one or more cesarean delivaries

Exclusion Criteria:

* Molar pregnancy.
* Fibroid uterus.
* Uterine anomalies.
* Coagulopathy.
* Medical disorder that contraindicate induction of abortion (e.g. heart failure).
* Previous attempts for induction of abortion in the current pregnancy.
* Allergy to misoprostol or letrozole.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-05 (Estimated); Primary Completion 2020-04-05 (Estimated); Study Completion 2020-04-10 (Estimated)

PRIMARY OUTCOMES:
induction to abortion time | 6 hours
  induction to abortion time
Incidence of complete miscarriage | 6 hours
  Incidence of complete miscarriage

SECONDARY OUTCOMES:
Need for surgical evacuation of the products of conception | 6 hours
  Need for surgical evacuation of the products of conception

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, Principal Investigator — Cairo University